CLINICAL TRIAL: NCT00905710
Title: Chromoendoscopy in Lynch Syndrome Patients
Brief Title: Chromoendoscopy to Decrease the Risk of Colorectal Neoplasia in Lynch Syndrome
Acronym: ChromoLynch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Leiden University Medical Center (Other); Free University Medical Center (Other); University Medical Center Nijmegen (Other); The Netherlands Cancer Institute (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jan J Koornstra, dr, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ChromoLynch
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Lynch Syndrome
Keywords: colorectal adenomas; colorectal cancer; Lynch syndrome; chromoendoscopy
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Conventional colonoscopy
- 2 (Experimental): Colonoscopy using chromoendoscopy
  Interventions: Procedure: Chromoendoscopy

INTERVENTIONS:
Procedure: Chromoendoscopy — Chromoendoscopy: spraying of the mucosa of the right colon with indigo-carmine
  Arms: 2

SUMMARY:
Lynch syndrome (LS), or hereditary nonpolyposis colorectal cancer (HNPCC), is a hereditary disorder predisposing for colorectal cancer. To reduce the risk of colorectal cancer, patients undergo colonoscopy every 1-2 years. Chromoendoscopy is relatively new technique which improves the detection of adenomas, the precursor lesions of colorectal cancer. The aim of this study is to determine whether chromoendoscopy, including polypectomy of all detected lesions, reduces the development of colorectal neoplasia and the need for colectomy in LS patients.

DETAILED DESCRIPTION:
Lynch syndrome (LS), or hereditary nonpolyposis colorectal cancer (HNPCC), is an autosomally dominantly inherited disorder that accounts for 1-2 % of colorectal cancer cases. LS is caused by germline genomic alterations in one of the mismatch repair (MMR) genes hMLH1, hMSH2, hMSH6 and hPMS2. The lifetime incidence of colorectal cancer is 20-75 % in these mutation carriers. Individuals with LS-associated colorectal cancer differ from those with sporadic disease in several ways: the tumours are diagnosed at an earlier age; the majority of tumours is located in the proximal colon; there is an increased risk of developing synchronous or metachronous colorectal cancers and the prognosis relatively favourable compared to sporadic cases. It is generally accepted that LS associated colorectal cancers develop along the adenoma-carcinoma sequence as in sporadic cases. There is evidence suggesting that the adenoma-carcinoma sequence is accelerated in LS patients as compared to the general population.

Colonoscopic screening and subsequent removal of polyps at a 3-year interval in asymptomatic at-risk members of LS families has shown to reduce the incidence of colorectal cancer and improve overall survival. However, within such an interval in surveillance programs, interval cancers have been observed. It is therefore currently recommended that MMR gene mutation carriers should be kept under surveillance by regular colonoscopy every 1-2 years beginning at the age of 20-25 or 5-10 years younger than the earliest affected family member.

LS adenomas are predominantly located in the proximal colon and frequently carry villous architecture and high-grade dysplasia, markers that are associated with an increased risk of developing colorectal cancer. Even in LS adenomas smaller than 5-7 mm in size, high-grade dysplasia can be encountered. Therefore, the identification of high-risk precursor lesions in LS is considered of paramount importance.

It is known that conventional colonoscopy has a certain miss rate for colorectal neoplasms, especially small adenomas. A few years ago, the technique of chromoendoscopy was introduced. Chromoendoscopy, in which one of various dyes are sprayed onto the colonic mucosa via a spray catheter passed through the working channel of the endoscope, offers detailed evaluation of the mucosal surface. Indigo carmine is a contrast stain that is not absorbed and does not react with the surface mucosa. In 2 large randomised controlled trials chromoendoscopy significantly increased the detection of small adenomas in the proximal colon as compared to conventional colonoscopy. Recently, 2 trials in LS patients revealed that chromoscopic endoscopy improved the detection of adenomas, particularly flat lesions, compared to conventional colonoscopy. Together, these data suggest that chromoendoscopy may improve detection rates of significant neoplastic colonic lesions in LS patients. However, the true value of chromoendoscopy in the management of LS patients remains to be demonstrated.

The aim of this study is to determine whether chromoendoscopy, including polypectomy of all detected lesions, reduces the development of colorectal neoplasia and the need for colectomy in LS patients at follow-up endoscopy.

The results of the study will indicate the value of chromoendoscopy in the management of LS patients and whether the technique should be implemented in current surveillance procedures.

ELIGIBILITY:
Inclusion Criteria:

* proven carrier of a MLH1, MSH2 or MSH6 mutation
* age between 20 and 70 years
* written informed consent

Exclusion Criteria:

* previous large bowel surgery
* psychological/physical conditions hampering compliance with the study protocol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoints of the study are the number of adenomas, advanced adenomas, carcinomas at baseline and the number of the number of adenomas, advanced adenomas, carcinomas and the number of patients requiring colectomy at 2-year follow-up. | 2 years

SECONDARY OUTCOMES:
The secondary endpoints of the study are the number of complications from colonoscopy at baseline and at 2-year follow-up. | baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan J Koornstra, MD PhD, Principal Investigator — University Medical Center Groningen, netherlands; Jan H Kleibeuker, MD PhD, Study Director — University Medical Center Groningen, Netherlands
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Stoffel EM, Turgeon DK, Stockwell DH, Normolle DP, Tuck MK, Marcon NE, Baron JA, Bresalier RS, Arber N, Ruffin MT, Syngal S, Brenner DE; Great Lakes New England Clinical Epidemiology and Validation Center of the Early Detection Research Network. Chromoendoscopy detects more adenomas than colonoscopy using intensive inspection without dye spraying. Cancer Prev Res (Phila). 2008 Dec;1(7):507-13. doi: 10.1158/1940-6207.CAPR-08-0096. PMID 19139000
- [Background] Huneburg R, Lammert F, Rabe C, Rahner N, Kahl P, Buttner R, Propping P, Sauerbruch T, Lamberti C. Chromocolonoscopy detects more adenomas than white light colonoscopy or narrow band imaging colonoscopy in hereditary nonpolyposis colorectal cancer screening. Endoscopy. 2009 Apr;41(4):316-22. doi: 10.1055/s-0028-1119628. Epub 2009 Apr 1. PMID 19340735
- [Derived] Haanstra JF, Dekker E, Cats A, Nagengast FM, Hardwick JC, Vanhoutvin SA, de Vos Tot Nederveen Cappel WH, Vasen HF, Kleibeuker JH, Koornstra JJ. Effect of chromoendoscopy in the proximal colon on colorectal neoplasia detection in Lynch syndrome: a multicenter randomized controlled trial. Gastrointest Endosc. 2019 Oct;90(4):624-632. doi: 10.1016/j.gie.2019.04.227. Epub 2019 Apr 24. PMID 31028782